CLINICAL TRIAL: NCT03002506
Title: Pharmacokinetics of Ceftolozane/Tazobactam in Patients With Burns
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Much slower recruitment than anticipated
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 070619
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Burns; Pharmacokinetics
Keywords: ceftolozane; tazobactam
MeSH Terms: conditions — Burns | interventions — ceftolozane, tazobactam drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ceftolozane/tazobactam (Experimental): One dose of 3 grams ceftolozane/tazobactam will be administered to each study participant.
  Interventions: Drug: Ceftolozane/tazobactam

INTERVENTIONS:
Drug: Ceftolozane/tazobactam — Single dose of 2 grams/1 gram intravenously administered over 60 minutes.
  Other Names: Zerbaxa

SUMMARY:
This study will help provide information about how patients with burn handle two antibiotics (ceftolozane and tazobactam) and use that information to guide dosing recommendations for these patients. The 12 patients who complete the study will receive a single dose of 3 grams ceftolozane/tazobactam intravenously. We will collect blood and urine samples to determine how much of each antibiotic is in the body and urine at various times over a 24 hour period. This information will be used with previously published information from microbiology laboratories to perform simulations that will provide recommendations on optimal dosing recommendations of these antibiotics in patients with burns.

DETAILED DESCRIPTION:
A single dose pharmacokinetic study of ceftolozane and tazobactam will be conducted in patients with burns at the Burn Center at University Medical Center. A total of 12 adults aged 18 to 80 years with >/= 20% percent total body surface area burned will be required to complete the study. A single intravenous dose of ceftolozane and tazobactam of 2 grams/1 gram will be administered over 60 minutes and whole blood will be obtained predose and at 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, and 24 hours following the start of infusion. Urine samples (5 ml) will be collected from a urine collection bag (if the patient has urinated) at the following timepoints: 0-0.5, 0.5-1, 1-2, 2-4, 4-8, 8-12, and 12-24 hours for analysis of ceftolozane and tazobactam content. Urine for collected during each time period will be measured to determine urine volume for urine clearance calculations. The volume of urine in the urine over the entire 24 hour period and an aliquot sent for analysis of urine creatinine content to determine the patient's 24 hour creatinine clearance.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, ages 18-80 years, of all racial and ethnic origins.
2. Non-English Spanish speakers will be included in the study.
3. We are recruiting 12 patients with thermal burn injuries (percent total body surface area burned >/= 20%). Patients will be at least five days from the date of the burn injury.
4. Patients will have central venous or arterial line access.
5. Patients will be already be receiving standard of care antimicrobial therapy for a suspected infection.

Exclusion Criteria:

1. Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of ceftolozane and tazobactam on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of ceftolozane and tazobactam, so that the pregnancy and post-partum state would be a confounding variable.
2. Abnormal liver function tests: transaminases >10 times upper limit of normal, Alkaline phosphatase >5 times upper limit of normal, total bilirubin >5 times upper limit of normal.
3. History of allergies to beta-lactam antibiotics.
4. Patients unwilling to comply with study procedures.
5. Current or previous participation within 28 days of enrollment in another research study that involves the use of medication, contrast, or any other compound that may alter blood count and/or blood chemistry (liver function, kidney function or electrolyte balance), unless waved by principal investigator (PI).
6. Donation of 450mL (one unit) of blood or more within 8 weeks (56 days) prior to study enrollment, unless waved by PI.
7. Creatinine clearance < 30 ml/min as estimated by the Cockcroft-Gault equation.
8. Patients who are receiving piperazillin/tazobactam or have received piperacillin/tazobactam within the past 48 hours.
9. Patients who are receiving vasopressors.
10. Patients with a total body weight < 60 kg or > 130 kg.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Hall, PharmD, Principal Investigator — Texas Tech University HSC
Locations (1):
- University Medical Center, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ceftolozane/Tazobactam
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants who provided informed consent and received ceftolozane/tazobactam.
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.67 (13.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Ceftolozane Clearnace
Description: Liters/hour (continuous values)
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: Liters per hour
Arm/Group | Ceftolozane/Tazobactam
Number analyzed (Participants) | 6
Liters per hour | 7.79 (2.30)

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Adverse events were to be reported if reported by the participant, healthcare team member, research team member, or lab documented.
Arm/Group | Ceftolozane/Tazobactam
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Single-dose pharmacokinetic study. No clinical outcomes to evaluate efficacy. No safety data provided by this study beyond a single dose in this population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT03002506/Prot_SAP_000.pdf